CLINICAL TRIAL: NCT01694810
Title: A Phase 1 Multiple Dose, Single-Center, Observer-Blind Parallel Group Study Evaluating Safety and Cutaneous Tolerability of NVN1000 Topical Gel in Healthy Volunteers
Brief Title: Cutaneous Tolerability and Safety of NVN1000 Topical Gel in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NI-AC002
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — berdazimer sodium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2% NVN1000 Topical Gel (Experimental): 2% NVN1000 Topical Gel once daily for 4 weeks
  Interventions: Drug: 2% NVN1000 Topical Gel
- 4% NVN1000 Topical Gel (Experimental): 4% NVN1000 4% Topical Gel once daily for 4 weeks
  Interventions: Drug: 4% NVN1000 Topical Gel
- Vehicle Topical Gel (Placebo Comparator): Vehicle Topical Gel once daily for 4 weeks
  Interventions: Drug: Vehicle Topical Gel
- 8% NVN1000 Topical Gel (Experimental): 8% NVN1000 8% Topical Gel applied once daily for 4 weeks
  Interventions: Drug: 8% NVN1000 Topical Gel

INTERVENTIONS:
Drug: 2% NVN1000 Topical Gel — 2% NVN1000 Topical Gel once daily for 4 weeks
  Other Names: NVN1000
  Arms: 2% NVN1000 Topical Gel
Drug: 4% NVN1000 Topical Gel — 4% NVN1000 4% Topical Gel applied once daily 4 weeks
  Other Names: NVN1000
  Arms: 4% NVN1000 Topical Gel
Drug: 8% NVN1000 Topical Gel — 8% NVN1000 Topical Gel applied once daily for 4 weeks
  Other Names: NVN1000
  Arms: 8% NVN1000 Topical Gel
Drug: Vehicle Topical Gel — Vehicle Topical Gel applied once daily
  Other Names: Vehicle
  Arms: Vehicle Topical Gel

SUMMARY:
The study will assess safety and tolerability of different doses of topical gel containing a new chemical entity, NVN1000, and the vehicle (gel without drug) applied to the face of healthy volunteers with high counts of Propionibacterium acnes. The test product will be applied once daily for 4 weeks. Exploratory measures include whether the topical product decreases the amount of a bacteria associated with acne (P. acnes).

DETAILED DESCRIPTION:
This is a single center, observer blinded, randomized, multiple dose study with 3 doses of NVN1000 and vehicle applied once daily for 4 weeks. There are 4 arms to the study (3 active and 1 vehicle).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers
* Age 18 or older
* High degree of fluorescence of facial skin under Wood's lamp

Exclusion Criteria:

* Acute or chronic skin disorders
* Use of topical or systemic antibiotics within 4 weeks of study
* Concomitant use of nitroglycerin or other nitric oxide donor drugs
* Females who are pregnant, planning pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Cutaneous tolerability Evaluation | 4 weeks
  Cutaneous tolerability evaluations to include erythema, scaling, dryness, puritus and burning/stinging using a 4-category scale with scores ranging from 0-3 (0=none, 1=mild, 2=moderate, 3 - severe).

SECONDARY OUTCOMES:
Safety Assessment | 4 weeks
  Comparison of adverse events between groups.
Safety Assessment | 4 weeks
  Change from baseline in HCT (L/L)
Safety Assessment | 4 weeks
  Change from baseline in HGB, MCHC (g/L)
Safety Assessment | 4 weeks
  Change from baseline in % methemoglobin (%)
Safety Assessment | 4 weeks
  Change from baseline in % Basophils (%)
Safety Assessment | 4 weeks
  Change from baseline in % Eosinophils (%)
Safety Assessment | 4 weeks
  Change from baseline in % Lymphocytes (%)
Safety Assessment | 4 weeks
  Change from baseline in MCH (pg)
Safety Assessment | 4 weeks
  Change from baseline in MCV, MPV (fL)
Safety Assessment | 4 weeks
  Change from baseline in % Monocytes (%)
Safety Assessment | 4 weeks
  Change from baseline in % Neutrophils (%)
Safety Assessment | 4 weeks
  Change from baseline in Platelet Count, WBC (10 ^ 9/L)
Safety Assessment | 4 weeks
  Change from baseline in % RDW (%)
Safety Assessment | 4 weeks
  Change from baseline in RBC (10 ^ 12/L)
Safety Assessment | 4 weeks
  Change from baseline in Albumin, Protein, Total (g/L)
Safety Assessment | 4 weeks
  Change from baseline in Alkaline Phosphatase, ALT, AST, (U/L)
Safety Assessment | 4 weeks
  Change from baseline in Bicarbonate, Bun, Calcium, Chloride, Glucose, Phosphorus, Potassium, Sodium (mmol/L)
Safety Assessment | 4 weeks
  Change from baseline in Bilirubin Direct, Bilirubin Total, Creatinine (umol/ L)

CONTACTS AND LOCATIONS:
Overall Officials: James J Leyden, MD, Principal Investigator — KGL, Inc.
Locations (1):
- KGL, Inc, Broomall, Pennsylvania, United States